CLINICAL TRIAL: NCT00336401
Title: Peri-Operative And Long-Term Cardioprotective Properties Of Sevoflurane In High Risk Patients Undergoing Non-Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Scott Beattie, Toronto General Hospital, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UHN REB 05-0011-B
Record Dates: First submitted 2006-06-08; First posted 2006-06-13 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2006-09

CONDITIONS: Non Cardiac Surgery
Keywords: anesthesia; non cardiac surgery; cardiac outcomes
MeSH Terms: interventions — Sevoflurane; Propofol

INTERVENTIONS:
Drug: Sevoflurane or Propofol

SUMMARY:
Non-cardiac surgery is associated with significant cardiac morbidity and mortality. Volatile anesthetics have a cardioprotective effects which results in preservation of left ventricular function and lower troponin I levels. Lower troponin release has been correlated with better long term event free survival in both cardiac and non cardiac surgery. A recently completed meta-analysis suggests that sevoflurane is a superior volatile agent. The evidence of a cardioprotective effect in non-cardiac surgery is lacking. Base on the current literature, we intend to evaluate the protective potential of sevoflurane versus propofol anesthesia in high risk patients undergoing elective non-cardiac procedures.

Hypothesis: The use of Sevoflurane as a general anesthetic reduces postoperative troponin release, the incidence of myocardial infarction and/or long term morbidity in patients at low to moderate risk of postoperative cardiac complications, who are undergoing noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

Any patient undergoing non-cardiac surgery is eligible if s/he: 1.) is ≥45 years old;2.) Has an expected length of stay ≥48 hours; AND3.) Fulfills any 2 of the six criteria for high cardiac risk as defined by the revised Cardiac Risk Index.(see details in protocol)4.) Informed consent

Exclusion criteria:A patient will be ineligible for this study if s/he:1) Prior adverse reaction to sevoflurane (MH patient) or propofol.2) Previous coronary artery bypass graft (CABG) surgery with complete revascularization in the preceding five years with no evidence of cardiac ischemia since the procedure; or3) Has concomitant life-threatening disease likely to limit life expectancy to <30 days. -

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-10; Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Beattie, MD, PhD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada